CLINICAL TRIAL: NCT00490308
Title: Blinded Randomised Trial About the Influence of Estradiol Supplementation During the Luteal in Patients Undergoing in Vitro Fertilization (IVF) Treatment
Brief Title: The Influence of Estradiol Supplementation During the Luteal in Patients Undergoing IVF Treatment
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 870/070
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2007-06-26 (Estimated); Status verified 2007-06

CONDITIONS: Infertility
Keywords: luteal; phase; estradiol; pregnancy; rate
MeSH Terms: conditions — Infertility | interventions — Therapeutics; Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Treatment with estradiol valerate

SUMMARY:
To evaluate whether treatment with Estradiol supplementation during the luteal phase improves IVF outcomes

Patients undergoing IVF treatment with controlled ovarian hyperstimulation using a GnRH analog will receive 4 mg estradiol valerate in the luteal phase.Patient's followup will include E2 progesterone and BHCG 14 days after embryo transfer and vaginal ultrasound on day 21 and 28 after embryo transfer

DETAILED DESCRIPTION:
The study will include Patients undergoing IVF treatment with controlled ovarian hyperstimulation using a daily GnRH analog in a long protocol,older then 18, .The women will be randomised to two groups.Both groups will be given vaginal tabs of natural micronized progesterone(Uterogestan)

The study group will be given oral estradiol Valerate 4 mg.Prior to treatment, each patient will be signed on informed concent.

Patients will be excluded if they are older than 40, have any systemic illnesses or a personal or family history of a thromboembolic event.

Follow up:

Verification of pregnancy status and hormonal profile will be carried out on day fourteen after embryo transfer by means of serum hCG,P and E2. clinical pregnancy will be defined as the presence of a gestational sac on ultrasonography on day 21 after embryo transfer and fetal heart will be evaluated on day 28

ELIGIBILITY:
Inclusion Criteria:

* Women treated for infertility with controlled ovarian hyperstimulation using daily GnRH agonist

Exclusion Criteria:

* Women younger then 18 or older then 40
* Women with systemic disease
* Women with a family or personal history of thromboembolic event

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-08; Study Completion 2008-08 (Estimated)

SECONDARY OUTCOMES:
E2 and progesterone levels

CONTACTS AND LOCATIONS:
Overall Officials: Rephael Ron-el, profesor, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Infertilty unit, Assaf-Harofeh Medical Center, Ẕerifin, Israel